CLINICAL TRIAL: NCT01818531
Title: Evaluation of Ultrasound-Guided Adductor Canal Blockade for Postoperative Analgesia Following Robotic Medial Unicompartmental Knee Replacement
Brief Title: Adductor Canal Block for Medial Compartment Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00023002
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Postoperative Analgesia; Medial Unicompartmental Knee Arthroplasty
Keywords: Partial knee replacement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adductor canal block (Experimental): Patients in this arm will receive an adductor canal block prior to undergoing a medial compartment knee arthroplasty.
  Interventions: Drug: Adductor canal block
- Lumbar plexus block (Active Comparator): Patients in this arm will receive a lumbar plexus block prior to undergoing a medial compartment knee arthroplasty.
  Interventions: Drug: Lumbar plexus block

INTERVENTIONS:
Drug: Adductor canal block
  Other Names: Saphenous nerve block
  Arms: Adductor canal block
Drug: Lumbar plexus block
  Arms: Lumbar plexus block

SUMMARY:
This study will evaluate the affects of a single injection ultrasound-guided adductor canal block for patients undergoing robotic-assisted (MAKOplasty) medial UKA (unicompartmental knee arthroplasty). Specifically, this study will compare the adequacy of postoperative analgesia provided by the adductor canal block with that provided by single injection lumbar plexus blockade. The working hypothesis is that the analgesia provided by the adductor canal block will be equivalent to the analgesia provided by the lumbar plexus block. The primary outcome will be a comparison of verbal numerical pain scores at rest and with movement over the first 24 hours following nerve blockade.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85
* Undergoing unilateral robotic-assisted (MAKOplasty) medial compartment knee arthroplasty at Wake Forest University Baptist Medical Center.
* Must give written informed consent for anesthesia including subarachnoid blockade and peripheral nerve blockade of both the lumbar plexus and adductor canal.
* Must consent to the performance of a sham block at the site to which they are not randomized.
* Must also be reliable to give accurate verbal pain scores postoperatively.

Exclusion Criteria:

* Contraindication to adductor canal blockade or lumbar plexus blockade (including significant coagulation abnormalities)
* History of opioid addiction or current chronic pain therapy for pain other than at the surgical site that is being treated with high-dose opioids (extended release opioids or > 40mg oxycodone equivalents per day)
* Allergy to study medications
* Failure to adequately place either the adductor canal or lumbar plexus blocks.
* Patients who decline or have a contraindication to subarachnoid blockade will also be excluded from the study.
* Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl S Henshaw, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Meek RM, Masri BA, Duncan CP. Minimally invasive unicompartmental knee replacement: rationale and correct indications. Orthop Clin North Am. 2004 Apr;35(2):191-200. doi: 10.1016/S0030-5898(03)00115-9. PMID 15062705
- [Background] Riddle DL, Jiranek WA, McGlynn FJ. Yearly incidence of unicompartmental knee arthroplasty in the United States. J Arthroplasty. 2008 Apr;23(3):408-12. doi: 10.1016/j.arth.2007.04.012. Epub 2007 Nov 26. PMID 18358380
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] GARDNER E. The innervation of the knee joint. Anat Rec. 1948 May;101(1):109-30. doi: 10.1002/ar.1091010111. No abstract available. PMID 18915634
- [Background] Davis JJ, Bond TS, Swenson JD. Adductor canal block: more than just the saphenous nerve? Reg Anesth Pain Med. 2009 Nov-Dec;34(6):618-9. doi: 10.1097/AAP.0b013e3181bfbf00. No abstract available. PMID 19901788
- [Background] Horner G, Dellon AL. Innervation of the human knee joint and implications for surgery. Clin Orthop Relat Res. 1994 Apr;(301):221-6. PMID 8156678
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Lund J, Jenstrup MT, Jaeger P, Sorensen AM, Dahl JB. Continuous adductor-canal-blockade for adjuvant post-operative analgesia after major knee surgery: preliminary results. Acta Anaesthesiol Scand. 2011 Jan;55(1):14-9. doi: 10.1111/j.1399-6576.2010.02333.x. Epub 2010 Oct 29. PMID 21039357
- [Background] Farrar JT, Berlin JA, Strom BL. Clinically important changes in acute pain outcome measures: a validation study. J Pain Symptom Manage. 2003 May;25(5):406-11. doi: 10.1016/s0885-3924(03)00162-3. PMID 12727037
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848

RESULTS

PARTICIPANT FLOW:
Groups:
- Adductor Canal Block: Patients in this arm will receive an adductor canal block prior to undergoing a medial compartment knee arthroplasty.
  Adductor canal block
- Lumbar Plexus Block: Patients in this arm will receive a lumbar plexus block prior to undergoing a medial compartment knee arthroplasty.
  Lumbar plexus block
Period: Overall Study
Arm/Group | Adductor Canal Block | Lumbar Plexus Block
Started | 75 | 75
Completed | 74 | 73
Not Completed | 1 | 2
Not completed — Withdrawn for case delay after block | 1 | 0
Not completed — Withdrawn for long-acting opioid patch | 0 | 1
Not completed — Withdrawn for failure to place block | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adductor Canal Block | Lumbar Plexus Block | Total
Number analyzed (Participants) | 74 | 73 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10.2) | 63 (10.5) | 63 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 39 | 72
  Male | 41 | 34 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 63 | 63 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Verbal Pain Scores at 6 Hours Post Nerve Blockade.
Description: Comparison of verbal numerical pain scores at rest and with movement 6 hours following nerve blockade. The score range is 0-10 with higher scores denoting worse outcomes.
Time Frame: 6 hours post block.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adductor Canal Block | Lumbar Plexus Block
Number analyzed (Participants) | 74 | 73
score on a scale
  rest | 1 (2) | 1.1 (2.2)
  movement | 1.6 (2.6) | 1.5 (2.8)

2. Secondary Outcome: Opioid Consumption
Description: Comparison of cumulative opioid consumption over 24 hour period between adductor canal block and lumbar plexus block.
Time Frame: 6, 12, 18, and 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Adductor Canal Block | Lumbar Plexus Block
Number analyzed (Participants) | 74 | 73
mg
  6 hours | 1.5 (4.5) | 2.5 (5.2)
  12 hours | 11 (14.3) | 10.3 (11.5)
  18 hours | 20.9 (26.8) | 20.7 (17.8)
  24 hours | 27.9 (38.4) | 32.1 (27.7)

3. Secondary Outcome: Time to First Analgesic
Description: Time to first analgesic between two groups: adductor canal block and lumbar plexus block.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Adductor Canal Block | Lumbar Plexus Block
Number analyzed (Participants) | 74 | 73
minutes | 601 (295) | 659 (366)

4. Secondary Outcome: Opioid Related Side Effects
Description: Occurrence of opioid related side effects (nausea, vomiting and pruritus) between two groups: adductor canal block and lumbar plexus block.
Time Frame: 6, 12, 18, and 24 hours
Measure: Number; unit: events
Arm/Group | Adductor Canal Block | Lumbar Plexus Block
Number analyzed (Participants) | 74 | 73
events
  Nausea 6 hours | 14 | 15
  Nausea 12 hours | 10 | 16
  Nausea 18 hours | 5 | 8
  Nausea 24 hours | 9 | 15
  Vomiting 6 hours | 6 | 8
  Vomiting 12 hours | 6 | 6
  Vomiting 18 hours | 2 | 3
  Vomiting 24 hours | 4 | 6
  Pruritus 6 hours | 11 | 3
  Pruritus 12 hours | 7 | 4
  Pruritus 18 hours | 5 | 5
  Pruritus 24 hours | 10 | 13

5. Secondary Outcome: Quadriceps Motor Strength
Description: Comparison of quadriceps motor strength at 6 hour post nerve block between two groups: adductor canal block and lumbar plexus block. The score range is 0-5, with higher scores denoting better outcomes.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adductor Canal Block | Lumbar Plexus Block
Number analyzed (Participants) | 74 | 73
units on a scale | 4 (1.1) | 2.5 (1.3)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Adductor Canal Block | Lumbar Plexus Block
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/73
Other Adverse Events (participants affected / at risk) | 38/74 | 43/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adductor Canal Block (N=74) | Lumbar Plexus Block (N=73)
Nausea (Gastrointestinal disorders) | 25 | 32
Vomitting (Gastrointestinal disorders) | 15 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes